CLINICAL TRIAL: NCT02135991
Title: Preparing to Run Effective Prevention
Acronym: PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R01AA022353 (NIH)
Record Dates: First submitted 2014-05-06; First posted 2014-05-12 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Implementation of Evidence Based Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Project CHOICE + Getting To Outcomes (Experimental): Boys and Girls Club sites will receive a) training and materials for Project CHOICE and b) training, ongoing technical assistance for two years, and materials for Getting To Outcomes
  Interventions: Behavioral: Getting To Outcomes; Behavioral: Project CHOICE
- Project CHOICE only (Active Comparator): Boys and Girls Club sites will receive a) training and materials for Project CHOICE
  Interventions: Behavioral: Project CHOICE

INTERVENTIONS:
Behavioral: Getting To Outcomes — These sites will receive written materials, training, and on site technical assistance to use the Getting To Outcomes process to implement Project CHOICE at their sites.
  Arms: Project CHOICE + Getting To Outcomes
Behavioral: Project CHOICE — Sites will receive standard training for Project CHOICE.

SUMMARY:
Young people can engage in a variety of negative behaviors-such as drug use, underage drinking, and premarital sex-that exact a high toll on local communities. These activities are often the target of community-based prevention efforts. Getting To Outcomes (GTO) is an approach that includes a toolkit, technical assistance, and training, organized around a 10-step process, that helps communities plan, implement, and evaluate the impact of their programs that attempt to prevent these negative behaviors. This study will examine the degree to which Getting To Outcomes helps Boys and Girls Clubs implement an evidence based drug prevention program.

DETAILED DESCRIPTION:
As a nation, the U.S. invests heavily in community-based organizations to conduct interventions, proven through research, to reduce the high rates of alcohol and drug use among teens. Much less is invested in helping communities implement these programs with quality. Although many evidence-based programs exist to address alcohol and drug use, communities face difficulty implementing them and achieving the same outcomes as researchers. This "gap" is because resources are limited, prevention is complex, and communities often lack the capacity-or the knowledge, attitudes, and skills-needed to implement "off the shelf" programs well. Common ways to bridge this gap, such as information dissemination, fail to change practice or outcomes at the local level in part because it does not sufficiently address capacity of community practitioners. Therefore, building a community's capacity is a method that could improve the quality of implementation and outcomes. Getting To Outcomes (GTO) is an implementation support intervention shown to improve the capacity of practitioners to conduct evidence-based programs, but its impact on fidelity and youth outcomes has not been studied. The study-Preparing to Run Effective Prevention (PREP)-will be a cluster randomized controlled trial using primary data from middle school youth (990) and program staff from 33 cooperating Boys and Girls Clubs sites (Sites) to assess how GTO impacts the fidelity, outcomes, and costs of an evidence-based program to prevent alcohol and drug use (Project CHOICE, PC). All 33 sites will receive training in PC. 16 Sites will conduct PC in a way typical of community-based organizations (PC only); 17 Sites will conduct PC augmented by GTO, comprised of training, onsite technical assistance, and a written GTO manual. The study will: (1) Assess the use of GTO and compare Sites' capacity between PC+GTO and PC only; (2) Compare PC fidelity between PC+GTO and PC only groups; (3) Compare alcohol and marijuana outcomes of middle-school youth in the PC+GTO (n=510) and PC only (n=480) groups; and (4) Assess the cost-effectiveness of GTO' impact. To address these aims we will collect data on the delivery and utilization of GTO (e.g., method of delivery, duration, topics); staff capacity to implement research-based interventions; observations of program delivery (fidelity monitoring); youth participants' use of, and attitudes towards, alcohol and marijuana via a survey at baseline and 3 and 6 months follow-up; and costs of both PC alone and PC+GTO. Analyses will examine differences between intervention (PC+GTO) and control (PC only) Sites' capacity, PC fidelity, outcomes, and costs over time, accounting for clustering within site. The PREP study could expand implementation research and serve as a model for how the government and other agencies support strong implementation of evidence-based programs in a wide array of domains. These outcomes are important to providing opportunities for youth to become healthy and productive adults.

ELIGIBILITY:
Youth participants

Inclusion Criteria:

Age 10-14 and attends a participating boys and girls club

Exclusion Criteria:

Younger than 10, older than 14, does not attend a participating boys and girls club

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 990 (Actual)
Dates: Start 2013-09; Primary Completion 2018-02 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Drug use | Baseline, 3 months, 6 months
  initiation and past month prevalence of alcohol use, marijuana use, perceptions of their friends' use of alcohol and marijuana, and resistance self-efficacy

SECONDARY OUTCOMES:
Fidelity | Each site will implement the 5 sessions of Project Choice twice (one time a year, for two years). In each year, we will collect fidelity data on two of the five sessions, for a total of 4 sessions rated over the two year period, for each site.
  (1) Adherence - local data collectors will rate how closely BGC staff adhered to the protocol as designed. (2) Dosage - BGC staff will record attendance of each participant (noting late arrivals/early leavers) and number minutes spent teaching each module. (3) Quality of delivery - Local data collectors will audio record visited sessions and send recordings to be rated by trained raters on the Motivational Interviewing Treatment Integrity Scale 3.1 (MITI).
Capacity | Annually for the first four years
  We will use the Capacity Interview to assess BGC staff capacity to conduct high-quality programming. Capacity ratings are made at the program level since programs operate as a unit. The ratings are made using a structured interview with key program personnel. The Capacity Interview has 14 items ("components") tied to each of the ten steps of the GTO model, averaging to a Total Score. Each component has seven responses, described with specific observable behaviors, ranging from "highly faithful" to "highly divergent" from ideal prevention practice.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Chinman, PhD, Principal Investigator — RAND
Locations (15):
- United States (15):
  - BGC of Buena Park, Buena Park, California
  - BGC of Burbank and Greater E Valley, Burbank, California
  - BGC of Carson, Carson, California
  - BGC of South Bay, Harbor City, California
  - BGC of East LA, Los Angeles, California
  - Challengers Boys and Girls Club, Los Angeles, California
  - Salesian BGC, Los Angeles, California
  - BGC of Santa Monica, Los Angeles, California
  - BGC of West Valley, Los Angeles, California
  - East Valley Boys and Girls Club, Los Angeles, California
  - BGC of Santa Ana, Los Angeles, California
  - BGC of LA Harbor, San Pedro, California
  - BGC Stanton, Stanton, California
  - BGC of Westminster, Westminster, California
  - BGC of Whittier, Whittier, California

REFERENCES:
- [Derived] Acosta J, Chinman M, Ebener PA, Malone PS, Cannon JS, D'Amico EJ. Sustaining an Evidence-Based Program Over Time: Moderators of Sustainability and the Role of the Getting to Outcomes(R) Implementation Support Intervention. Prev Sci. 2020 Aug;21(6):807-819. doi: 10.1007/s11121-020-01118-2. PMID 32323166
- [Derived] Herman PM, Chinman M, Cannon J, Ebener P, Malone PS, Acosta J, D'Amico EJ. Cost Analysis of a Randomized Trial of Getting to Outcomes Implementation Support of CHOICE in Boys and Girls Clubs in Southern California. Prev Sci. 2020 Feb;21(2):245-255. doi: 10.1007/s11121-019-01082-6. PMID 31865544
- [Derived] Cannon JS, Gilbert M, Ebener P, Malone PS, Reardon CM, Acosta J, Chinman M. Influence of an Implementation Support Intervention on Barriers and Facilitators to Delivery of a Substance Use Prevention Program. Prev Sci. 2019 Nov;20(8):1200-1210. doi: 10.1007/s11121-019-01037-x. PMID 31473932
- [Derived] Chinman M, Ebener P, Malone PS, Cannon J, D'Amico EJ, Acosta J. Testing implementation support for evidence-based programs in community settings: a replication cluster-randomized trial of Getting To Outcomes(R). Implement Sci. 2018 Oct 22;13(1):131. doi: 10.1186/s13012-018-0825-7. PMID 30348227